CLINICAL TRIAL: NCT06519032
Title: Development and Evaluation of Rapid Bacterial Species Identification for Acid-Fast Bacilli Smear Using Image Analysis AI
Status: Recruiting | Type: Observational
Sponsor: GramEye (Industry)
Collaborators: Osaka University (Other); Keio University (Other); Fukujuji Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: GE004
Record Dates: First submitted 2024-07-12; First posted 2024-07-25 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Bacterial Infections
MeSH Terms: conditions — Bacterial Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Sputum and other specimen used for microbiologic testing
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to develop AI that detects and classifies Acid-Fast Bacilli from microscope images using anonymized and fixed glass slides.

ELIGIBILITY:
Inclusion Criteria:

* Patients in whom acid-fast bacilli(AFB) smear test was ordered

Exclusion Criteria:

* No exclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Specimens for microbiological testing, such as acid-fast bacilli(AFB) smear test , ordered at the hospital.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2023-09-20 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Rate of concordance between AI-estimated results with actual culture results regarding the presence or absence of acid-fast bacteria | Day1
  Evaluate the difference between actual medical record reports(such as culture results) and AI-estimated results regarding the presence or absence of acid-fast bacteria

CONTACTS AND LOCATIONS:
Overall Officials: Satoshi Kutsuna, PhD,MD, Study Director — Osaka University Medical Hospital
Locations (1):
- Osaka University Hospital, Suita, Osaka, Japan